CLINICAL TRIAL: NCT06386458
Title: A Prospective, Multicenter, Randomized Controlled, Non-inferiority Clinical Study Evaluating the Safety and Efficacy of the AThrough Radiofrequency Transseptal Puncture System in Atrial Septal Puncture.
Brief Title: Assessing AThrough Radiofrequency Transseptal Puncture System for Left Atrial Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou NOYA MedTech Co. Ltm. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-01
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Heart Diseases; Atrial Fibrillation
MeSH Terms: conditions — Heart Diseases; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency transseptal puncture needle (Experimental): Utilizing Radiofrequency transseptal puncture system for left atrial access
  Interventions: Device: AThrough radiofrequency transseptal puncture system
- Traditional mechanical transseptal puncture needle (Active Comparator): Utilizing Traditional mechanical transseptal puncture needle for left atrial access
  Interventions: Device: Traditional mechanical transseptal puncture needle

INTERVENTIONS:
Device: AThrough radiofrequency transseptal puncture system — Utilizing AThrough radiofrequency transseptal puncture system for left atrial access
  Arms: Radiofrequency transseptal puncture needle
Device: Traditional mechanical transseptal puncture needle — Utilizing Traditional mechanical transseptal puncture needle for left atrial access
  Arms: Traditional mechanical transseptal puncture needle

SUMMARY:
This study is a prospective, multicenter, randomized controlled trial with a non-inferiority design. Participants are patients scheduled for atrial septal puncture. After signing informed consent, subjects will be randomly assigned to either the radiofrequency transseptal puncture system group (referred to as the trial group) or the traditional mechanical transseptal puncture system group (referred to as the control group). All participants will undergo immediate postoperative and discharge clinical follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥ 18 years;
2. Subjects scheduled to undergo cardiology interventional treatment via the transseptal puncture route;
3. Subjects have been informed about the nature of the study, understand the purpose of the clinical trial, and voluntarily participate and sign the informed consent form.

Exclusion Criteria:

1. Echocardiogram indicates the presence of intracardiac masses, thrombi, or vegetations; left atrial myxoma;
2. Subjects with an atrial septal defect occluder or atrial septal patch implant;
3. Hemorrhagic disease or coagulopathy; or contraindications to antithrombotic medication treatment;
4. Acute myocardial infarction occurred within the last 4 weeks;
5. End-stage heart failure (ACC/AHA stage D); post-heart transplant; or awaiting heart transplant;
6. Pregnant or breastfeeding women;
7. Acute systemic infection or sepsis;
8. Participation in any drug and/or medical device clinical trial within the last month;
9. Researchers judge the patient's compliance to be poor, unable to complete the study as required; or other situations deemed by the researchers as making the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Transseptal puncture success rate. | Intraprocedural assessment
  Defined as successfully completing the puncture in the atrial septum and establishing a pathway from the right atrium to the left atrium (with the sheath entering the left atrium) using the transseptal puncture system

SECONDARY OUTCOMES:
Initial transseptal puncture success rate. | Intraprocedural assessment
  Defined as the period from the introduction of the transseptal puncture system into the femoral vein to the entry of transseptal sheath into the left atrium.
Time required to successfully complete the transseptal puncture. | Intraprocedural assessment
  Defined as the time from when the transseptal puncture system is introduced into the femoral vein to when the transseptal sheath enters the left atrium.
Number of attempts needed to successfully complete the transseptal puncture. | Intraprocedural assessment
  During the transseptal puncture process, if the transseptal puncture system needs to be readjusted upwards and repositioned for oval fossa puncture, each readjustment should count as an additional attempt.
Ratio of atrial septal puncture failures that cross over to the opposite group. | Intraprocedural assessment
  Ratio of atrial septal puncture failures that cross over to the opposite group;

CONTACTS AND LOCATIONS:
Overall Officials: Wei Sun, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (4):
- China (4):
  - The 7th People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang